CLINICAL TRIAL: NCT07290361
Title: Stratified Targeted Engagement From Primary Care to Physical Therapy (STEPPT): A Pragmatic Stepped Wedge Cluster Randomized Trial
Brief Title: Stratified Targeted Engagement From Primary Care to Physical Therapy (STEPPT)
Acronym: STEPPT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Family Health Centers of San Diego (Other)
Responsible Party: Principal Investigator, Katrina Monroe, PT, PhD, San Diego State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: HS-2023-0122; R01MD018937 (NIH)
Record Dates: First submitted 2025-12-14; First posted 2025-12-18 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Low Back Pain; Neck Pain
Keywords: Physical therapy; Rehabilitation; Hispanic; Heatlh Services; Healthcare utilization; Federally Qualified Health Center
MeSH Terms: conditions — Low Back Pain; Neck Pain | interventions — Nurses

STUDY DESIGN:
Intervention Model Description: The STEPPT study will use a hybrid type 1, pragmatic stepped wedge cluster randomized trial (SW-CRT) design to evaluate implementation and effectiveness of a multi-level intervention aimed at improving rates of physical therapy referral and adherence among Hispanic patients with spine pain at a Federally Qualified Health Center. The unit of randomization is clinics. Outcomes will be assessed at the participant level.
Masking Description: The STEPPT trial will use single blind masking in which patients will remain blind to the study purpose and alternate care pathways (STEPPT Care vs. Usual Care) throughout the trial. Providers and clinic staff cannot be blinded due to the nature of the intervention (i.e., providers and staff require training to administer STEPPT and implement workflow changes). The order of cross-over from Usual Care to STEPPT will be concealed from investigators, providers, and staff until one month prior to each step in the SW-CRT. At this time, the statistician will communicate the clinics that have been randomly assigned to cross over to the FQHC Research Manager who will then initiate training activities which will unblind providers and staff. Primary and secondary outcomes will be assessed using automated algorithms applied to electronic health record (EHR) data to minimize bias. Investigators, providers, and staff will have access to these data for feedback and quality improvement purposes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STEPPT Care Pathway (Experimental): The STEPPT Care Pathway is a multi-level intervention designed to improve physical therapy (PT) referral and adherence among Hispanic patients with spine pain in Federally Qualified Health Center. STEPPT includes: 1) provider training and feedback through brief in-service education on guideline-based referral and culturally responsive communication about the benefits of PT for spine pain, 2) delivery of culturally tailored patient education materials in English and Spanish via print, video, and digital platforms, and 3) enhanced care navigation by bilingual Patient Health Navigators who provide personalized outreach, barrier mitigation, and scheduling support. System-level enhancements include automated electronic health record tools for patient identification, registry tracking, and delivery of education materials to ensure timely referral and engagement in PT services.
  Interventions: Behavioral: Engagement of clinic leadership (System Intervention - STEPPT); Behavioral: Patient Registry (System Intervention - STEPPT); Behavioral: Delivery of Patient Education Materials (System Intervention - STEPPT); Behavioral: Patient Health Navigator Training (System Intervention - STEPPT); Behavioral: Care Navigation (System Intervention - STEPPT); Behavioral: Care navigation audit and feedback (System Intervention - STEPPT); Behavioral: Primary Care Provider training (Provider Intervention - STEPPT); Behavioral: Nurse/Medical Assistant Training (Provider Intervention - STEPPT); Behavioral: Provider feedback on PT referral and adherence (Provider Intervention - STEPPT); Behavioral: Patient education on spine pain condition (Patient Intervention - STEPPT); Behavioral: Patient Education on Physical Referral by Providers (Patient Intervention - STEPPT); Behavioral: Electronic Patient Education on Physical Therapy Referral (Patient Intervention - STEPPT); Behavioral: Patient education on physical therapy referral by Patient Health Navigator (Patient Intervention - STEPPT); Behavioral: Monitoring of PT referral and adherence rates (System Intervention - STEPPT)
- Usual Care Pathway (Control) (Active Comparator): The Usual Care Arm involves the current institutional standard of referral and scheduling processes. If a patient is referred to physical therapy, a centralized Referral Specialist verifies insurance and attempts to schedule the evaluation. No provider/staff training, culturally tailored patient education, or enhanced care navigation is provided beyond the current standard of care.
  Interventions: Behavioral: Engagement of clinic leadership (System Intervention - Usual Care); Behavioral: Delivery of Patient Education Materials (System Intervention - Usual Care); Behavioral: Referral Specialist Training (System Intervention - Usual Care); Behavioral: Patient education on spine pain condition (Patient Intervention - Usual Care); Behavioral: Patient Education on Physical Referral by Providers (Patient Intervention - Usual Care); Behavioral: Patient education on physical therapy referral by Referral Specialist (Patient Intervention - Usual Care); Behavioral: Care Navigation (System Intervention - Usual Care); Behavioral: Monitoring of PT referral and adherence rates (System intervention - Usual Care)

INTERVENTIONS:
Behavioral: Engagement of clinic leadership (System Intervention - Usual Care) — No engagement of clinic leadership in promotion or monitoring of PT referral patterns among providers or PT adherence patterns among patients
  Arms: Usual Care Pathway (Control)
Behavioral: Engagement of clinic leadership (System Intervention - STEPPT) — Clinic Directors and Charge Nurses engage in STEPPT onboarding meeting with STEPPT Project Manager to discuss STEPPT objectives, procedures, and need for local adaptations. Medical leaders champion provider training and facilitate change in practice patterns through regularly scheduled review of trends in PT referral and adherence patterns with STEPPT Project Manager.
  Arms: STEPPT Care Pathway
Behavioral: Patient Registry (System Intervention - STEPPT) — Patients referred to physical therapy for spine pain are stratified by ethnicity. Hispanic patients are added to STEPPT Patient Registry to facilitate targeted engagement of an underserved population known to have low rates of adherence for physical therapy referrals.
  Arms: STEPPT Care Pathway
Behavioral: Delivery of Patient Education Materials (System Intervention - Usual Care) — Neck or back pain fact sheet may be manually ordered in the printed after visit summary at the discretion of the primary care physician. No automated systems for delivery of patient education materials on spine pain or physical therapy referral.
  Arms: Usual Care Pathway (Control)
Behavioral: Delivery of Patient Education Materials (System Intervention - STEPPT) — Automated delivery systems for patient education materials include:
  * Auto-order for culturally tailored neck or back pain fact sheet, general PT fact sheet, and postural exercise fact sheet printed in the AVS for all Hispanic patients with a new or existing spine pain problem
  * Auto-order for text message with links to culturally tailored PT referral fact sheet and video upon referral to PT for spine pain
  * Auto-order for culturally tailored neck or back pain fact sheet, general PT fact sheet, postural exercise fact sheet, PT referral fact sheet, and video added to the patient portal upon referral to PT for spine pain
  Arms: STEPPT Care Pathway
Behavioral: Referral Specialist Training (System Intervention - Usual Care) — Referral Specialists trained in system-wide procedures for processing referrals, calling patients, and scheduling appointments for specialty services. Physical therapy referrals processed by a dedicated team of Physical Rehabilitation Services Referral Specialists.
  Arms: Usual Care Pathway (Control)
Behavioral: Patient Health Navigator Training (System Intervention - STEPPT) — Patient Health Navigators (PHNs) trained in system-wide procedures for processing referrals, calling patients, and scheduling appointments for specialty services. Additional training on patient communication and enhanced care navigation is provided to address cultural factors, individual barriers, and risk factors for non-adherence. Physical therapy referrals processed by a specially trained team of Physical Rehabilitation Services PHNs.
  Arms: STEPPT Care Pathway
Behavioral: Care Navigation (System Intervention - STEPPT) — Upon referral to PT and verification of insurance coverage, patients receive a system-generated auto-call to schedule the PT evaluation followed by up to 3 phone contact attempts by a Patient Health Navigator (PHN) to 1) deliver enhanced care navigation, and 2) schedule PT evaluation. Prior to scheduling, PHN delivers semi-scripted enhanced care navigation (ECN) with mandatory components:
  * Summarize benefits of PT
  * Emphasize importance of attending PT even if prescribed medication for temporary pain relief
  * Confirm patient received and reviewed educational materials. Resend materials, if needed
  * Address privacy concerns, if present
  * Address risk factors for PT non-adherence, if present: scheduling, cost, transportation barriers
  * Address other questions or concerns
  * Schedule the PT evaluation
  * Repeat appointment details and provide PHN contact information for additional questions
  Arms: STEPPT Care Pathway
Behavioral: Care navigation audit and feedback (System Intervention - STEPPT) — Audits of fidelity to enhanced care navigation protocol using self-report checklists and review of recorded phone calls are discussed monthly with PHNs to facilitate competent and consistent delivery of enhanced care navigation for patients in STEPPT registry.
  Arms: STEPPT Care Pathway
Behavioral: Primary Care Provider training (Provider Intervention - STEPPT) — PCPs attend training with Physical Rehabilitation Services site manager on the following topics:
  * STEPPT objectives, procedures, and patient education materials
  * Referral and adherence rates for PT among Hispanic patients at FQHC clinics
  * Benefits of PT referral for patients with new and existing spine pain problems
  * Culturally responsive strategies to improve patient engagement in PT services (e.g., explanation of how PT can improve family and social role functioning)
  Arms: STEPPT Care Pathway
Behavioral: Nurse/Medical Assistant Training (Provider Intervention - STEPPT) — Nurses and MAs attend training with Physical Rehabilitation Services site manager on the following topics:
  * STEPPT objectives, procedures, and patient education materials
  * Referral and adherence rates for PT among Hispanic patients at FQHC clinics
  * Benefits of PT referral for patients with new and existing spine pain problems
  * Culturally responsive strategies to improve patient engagement in PT services (e.g., explanation of the FQHC referral process)
  Arms: STEPPT Care Pathway
Behavioral: Provider feedback on PT referral and adherence (Provider Intervention - STEPPT) — Trends in PT referral and adherence rates, stratified by ethnicity, are reviewed biannually at "Provider Huddles" along with suggestions for improvement as needed.
  Arms: STEPPT Care Pathway
Behavioral: Patient education on spine pain condition (Patient Intervention - Usual Care) — Verbal patient education on etiology, treatment, and prognosis for spine pain may be provided at the discretion of Primary Care Physician. Back Pain or Neck Pain Fact Sheet may be ordered in the printed After Visit Summary at the discretion of Primary Care Physician. Back Pain/Neck Pain Factsheet summarizes current evidence on etiology, prognosis, and treatment (medical and self-management) for back or neck pain. [Available in English or Spanish language]
  Arms: Usual Care Pathway (Control)
Behavioral: Patient education on spine pain condition (Patient Intervention - STEPPT) — Verbal patient education on etiology, treatment, and prognosis for spine pain may be provided at the discretion of Primary Care Physician. Patient education materials auto-ordered in the printed After Visit Summary for all patients with a new or existing spine pain problem on the electronic health record Problem List. STEPPT patient education materials include: (1) Back Pain or Neck Pain Facts, a culturally tailored factsheet summarizing current evidence on etiology, prognosis, and treatment (medical and self-management) for back or neck pain, (2) Physical Therapy Fact Sheet, culturally tailored information describing physical therapy evaluation and treatment options for pain with a QR code linking to a Physical Therapy Education Video, (3) Posture Exercises, culturally tailored instructions for standing posture, seated posture, and supine diaphragmatic breathing. [All patient education materials available in English or Spanish language]
  Arms: STEPPT Care Pathway
Behavioral: Patient Education on Physical Referral by Providers (Patient Intervention - Usual Care) — Verbal patient education on physical therapy referral may be provided at the discretion of Primary Care Physician, Nurse, and/or Medical Assistant at index encounter. Patients are notified of referral for physical therapy consultation in the printed After Visit Summary. No written instructions on physical therapy referral process are provided.
  Arms: Usual Care Pathway (Control)
Behavioral: Patient Education on Physical Referral by Providers (Patient Intervention - STEPPT) — Following training in best practices, primary care providers encouraged to provide culturally responsive patient education on benefits of PT for spine pain at index encounter. Nurses and medical assistants encouraged to review printed patient education materials on benefits of PT and institutional referral process. Patients are notified of referral for physical therapy consultation in the printed After Visit Summary at index encounter.
  Arms: STEPPT Care Pathway
Behavioral: Electronic Patient Education on Physical Therapy Referral (Patient Intervention - STEPPT) — Patient receives auto-email from patient portal and auto-text message with links to electronic patient education materials upon being referred to PT:
  * Physical Therapy Referral Information - Culturally tailored information highlighting the importance of attending PT, resources to support regular attendance, and instructions for scheduling and preparing for the PT evaluation. [Eng/Span]
  * Physical Therapy Education Video - Culturally tailored video showing how to schedule and attend the PT evaluation with testimonials from former FQHC patients highlighting benefits of PT for spine pain. [Eng/Span]
  Arms: STEPPT Care Pathway
Behavioral: Patient education on physical therapy referral by Referral Specialist (Patient Intervention - Usual Care) — Verbal patient education on physical therapy referral may be provided at the discretion of the Referral Specialist when scheduling the physical therapy consultation.
  Arms: Usual Care Pathway (Control)
Behavioral: Patient education on physical therapy referral by Patient Health Navigator (Patient Intervention - STEPPT) — Culturally responsive, semi-scripted patient education on benefits of physical therapy and logistics of physical therapy appointments provided verbally by a Patient Health Navigator (PHN) when scheduling the physical therapy consultation. PHN identifies and helps mitigate individual barriers for attending physical therapy appointments.
  Arms: STEPPT Care Pathway
Behavioral: Care Navigation (System Intervention - Usual Care) — Upon PT referral and verification of insurance coverage, patient receives up to 2 system-generated auto-calls to schedule PT evaluation. If no contact is made after 30 days, a system-generated letter is sent by mail requesting the patient call a centralized Referral Specialist to schedule the PT evaluation. Additional care navigation services may be provided at the discretion of the Referral Specialist.
  Arms: Usual Care Pathway (Control)
Behavioral: Monitoring of PT referral and adherence rates (System Intervention - STEPPT) — Automated EHR analysis monitors daily PT referral and adherence rates for spine pain. PowerBI custom graphical interface with monthly trends in PT referral and adherence rates, stratified by ethnicity, are reviewed biannually by Vice President of Specialty Services, Physical Rehabilitation Services site manager, medical leadership, and providers.
  Arms: STEPPT Care Pathway
Behavioral: Monitoring of PT referral and adherence rates (System intervention - Usual Care) — PT referral and adherence rates monitored as needed by Vice President of Specialty Services.
  Arms: Usual Care Pathway (Control)

SUMMARY:
The goal of this clinical trial is to learn if a health system intervention called "Stratified Targeted Engagement from Primary Care to Physical Therapy (STEPPT)" can improve how often doctors refer Hispanic patients with spine pain to physical therapy (referral rate) and how often patients attend physical therapy after being referred (adherence rate). The main questions this study aims to answer are 1) does STEPPT improve physical therapy referral and adherence rates compared to usual care for Hispanic patients with spine pain who seek care in a Federally Qualified Health Center (FQHC) serving low income communities, and 2) how consistently do FQHC providers and staff deliver STEPPT to patients who may benefit? STEPPT will train doctors and other health care providers to educate participants on the benefits of physical therapy for spine pain and participants will receive culturally tailored handouts and videos to teach them about their spine pain and what to expect in physical therapy. Patients will also receive personalized assistance to schedule their physical therapy appointment and address potential barriers for attending the appointment.

DETAILED DESCRIPTION:
This study will examine the implementation and effectiveness of STEPPT for improving access and engagement of Hispanic patients with spine pain in physical therapy (PT) services at a Federally Qualified Health Center (FQHC) serving low-income communities near the United States-Mexico border. A pragmatic hybrid type I stepped wedge cluster randomized trial (SW-CRT) will be conducted to examine the effectiveness of STEPPT for increasing rates of PT referral and adherence as a primary aim. The study will also explore implementation outcomes to better understand the context of enacting a targeted intervention to engage medically underserved populations as a secondary aim. Nine FQHC Primary Care clinics (clusters) will be randomized to three implementation steps, with three clinics allocated per step, using a covariate-constrained randomization approach. To minimize imbalance between steps, allocation of clinics will be balanced with respect to clinic size and historical rates of PT referral and adherence in the year prior to allocation. For each candidate allocation, an imbalance score summarizing differences across steps will be calculated and the randomization procedure will be repeated to identify the allocation yielding the smallest overall imbalance score as the final stepped-wedge assignment. The three steps will transition from Usual Care (control) to STEPPT (intervention) at 6-month intervals. A 6-month baseline period of Usual Care for all clinics will precede the first date of cross over into STEPPT. Implementation and effectiveness outcomes will be assessed at 6-month intervals throughout the trial.

ELIGIBILITY:
Inclusion Criteria

* 18 years or older.
* Identify as either Hispanic or Non-Hispanic ethnicity, inclusive of all races.
* Seeking care for spine pain at an Adult or Adult Walk-in primary care clinic within the participating Federally Qualified Health Center (FQHC).
* New or existing spine pain problem: A new spine pain problem is defined by a new ICD code for neck or back pain added to the problem list during a visit with a primary care physician. An existing spine pain problem is defined by an existing ICD code for neck or back pain on the problem list that is associated with a physician referral for any service during the visit related to the neck or back pain problem.
* Signed a broad consent for the use of de-identified health information for research at the participating FQHC.

Exclusion Criteria:

* Spine pain associated with a non-musculoskeletal etiology (e.g., infection, cancer, urological disorders, pregnancy, etc.)
* Patients requiring urgent medical intervention (e.g., fracture, cauda equina syndrome, etc)
* Active physical therapy referral for spine pain at the time of the index encounter.
* Previously referred to physical therapy through the STEPPT Care Pathway.
* Physical therapy referrals external to the FQHC will be excluded from the analysis of physical therapy adherence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17587 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Physical Therapy Referral | Patient level: 3-months after index PCP encounter; Clinic level: 6-, 12-, 18-, and 24-months after start of trial
  Proportion of enrolled patients who receive an internal or external referral to physical therapy following Primary Care Provider (PCP) index encounter for a new or existing episode of spine pain.
Physical Therapy Adherence | Patient level: 6-months after index physical therapy referral; Clinic level: 6-, 12-, 18-, and 24-months after start of trial
  Proportion of enrolled patients who complete a physical therapy evaluation at the Federally Qualified Health Center following an internal referral to physical therapy for a new or existing episode of spine pain.

SECONDARY OUTCOMES:
Maintenance Physical Therapy Referral | Patient level: 3-months after index PCP encounter; Clinic level: 30-months after start of trial
  Proportion of enrolled patients who receive an internal or external referral to PT following Primary Care Provider (PCP) index encounter for a new or existing episode of spine pain during the maintenance phase.
Maintenance Physical Therapy Adherence | Patient level: 6-months after index physical therapy referral; Clinic level: 30-months after start of trial
  Proportion of enrolled patients who complete a physical therapy evaluation at the Federally Qualified Health Center following an internal referral to physical therapy for a new or existing episode of spine pain during the maintenance phase.
Patient age | Upon enrollment
  Patient age in years recorded in electronic health record
Patient sex | Upon enrollment
  Patient sex at birth recorded in electronic health record
Patient race | Upon enrollment
  Patient race recorded in electronic health record
Patient ethnicity | Upon enrollment
  Patient ethnicity recorded in electronic health record
Patient birth place | Upon enrollment
  Patient country of birth recorded in electronic health record
Patient education | Upon enrollment
  Patient highest level of education recorded in electronic health record
Patient employment | Upon enrollment
  Patient employment status recorded in electronic health record
Patient relationship status | Upon enrollment
  Patient relationship status (e.g., married, divorced, etc.) recorded in electronic health record
Patient neighborhood status | Upon enrollment
  Neighborhood healthy places index (HPI) score based on patient zipcode
Patient food insecurity | Upon enrollment
  Patient food insecurity status based on PREPAR questionnaire recorded in electronic health record
Patient transportation status | Upon enrollment
  Patient transportation status based on PRAPARE questionnaire recorded in electronic health record
Patient insurance | Upon enrollment
  Patient insurance status (federal, private, uninsured, etc.) recorded in electronic health record
Patient language | Upon enrollment
  Patient preferred language recorded in electronic health record
Patient interpreter | Upon enrollment
  Patient request for interpreter during primary care visit recorded in electronic health record
Index clinic | Upon enrollment
  Name of Federally Qualified Health Center clinic at which index encounter for spine pain occurred recorded in electronic health record
Spine pain region | Upon enrollment
  Region of spine pain (neck, low back, both) recorded in electronic health record at index encounter
Spine pain acuity | Upon enrollment
  New or existing spine pain problem recorded in electronic health record at index encounter
Patient comorbidity | Upon enrollment
  Functional comorbidity index recorded in electronic health record
Patient existing prescriptions | Upon enrollment
  Type and number of existing prescriptions recorded in electronic health record at index encounter
Patient new prescriptions | Upon enrollment
  Type and number of new prescriptions recorded in electronic health record at index encounter
Patient referrals | Upon enrollment
  Type and number of specialty referrals recorded in electronic health record at index encounter
Clinic size | Upon crossover to STEPPT
  Number of spine pain encounters during baseline period for each participating primary care clinic
Clinic location | Upon crossover to STEPPT
  Geographic location of each participating primary care clinic
Clinic PT Services | Upon crossover to STEPPT
  Availability of onsite physical therapy services for each participating primary care clinic
Provider age | 6-, 12-, 18-, 24-, and 30-months after start of trial
  Ages of primary care providers employed at each participating clinic recorded in clinic operations records
Provider sex | 6-, 12-, 18-, 24-, and 30-months after start of trial
  Sex of primary care providers employed at each participating clinic recorded in clinic operations records
Provider race | 6-, 12-, 18-, 24-, and 30-months after start of trial
  Races of primary care providers employed at each participating clinic recorded in clinic operations records
Provider ethnicity | 6-, 12-, 18-, 24-, and 30-months after start of trial
  Ethnicities of primary care providers employed at each participating clinic recorded in clinic operations records
Provider education | 6-, 12-, 18-, 24-, and 30-months after start of trial
  Highest clinical degrees for primary care providers employed at participating clinics recorded in clinic operations records
Provider specialty | 6-, 12-, 18-, 24-, and 30-months after start of trial
  Types of clinical specialties for primary care providers employed at each participating clinic recorded in clinic operations records
Provider experience | 6-, 12-, 18-, 24-, and 30-months after start of trial
  Time elapsed between date of highest clinical degree for primary care providers at each participating clinic and date of index encounter
Duration of provider employment | 6-, 12-, 18-, 24-, and 30-months after start of trial
  Duration of employment at federally qualified health center for primary care providers at each participating clinic recorded in clinical operations records
PCP frequency of PT education | Prior to training, 6-months after crossover to STEPPT
  Primary care physician self-reported frequency of educating patients with spine pain about the benefits of physical therapy (never, rarely, sometimes, often, always)
PCP qualitative interviews | 3-months after cross over to STEPPT
  Qualitative interviews with primary care providers to assess motivations, barriers, and facilitators for any changes made in the rate of physical therapy referral and the frequency, content, and approach for patient education on benefits of physical therapy
Allied provider frequency of PT education | Prior to training, 6-months after crossover to STEPPT
  Nurse and Medical Assistant self-reported frequency of educating patients about the benefits of physical therapy and referral process (never, rarely, sometimes, often, always)
Allied provider qualitative interviews | 3-months after cross over to STEPPT
  Qualitative interviews with nurses and medical assistants to assess motivations, barriers, and facilitators for any changes made in the rate of physical therapy referral and the frequency, content, and approach for patient education on benefits of physical therapy
Training Involvement Rating Scale (IRS) score | 6-, 12-, 18-months after start of trial
  Scale ranging from 0-15 points quantifies unsatisfactory (0-5 points), moderate (6-10 points) and satisfactory (11-15 points) involvement of clinic staff in STEPPT trainings. IRS score assesses the following training domains: 1) clinic administrator orientation, 2) primary care physician orientation, 3) Nurse/Medical Assistant orientation, 4) Review of progress reports, 5) ECN training and audit reviews
ECN contact attempts | 12-, 18-, 24-, and 30-months after start of trial
  Number of enhanced care navigation call attempts prior to scheduling first physical therapy appointment
ECN completed contacts | 12-, 18-, 24-, and 30-months after start of trial
  Proportion of Hispanic patients referred to physical therapy who were able to be contacted by patient health navigator, regardless of whether enhanced care navigation was delivered
ECN delivery | 12-, 18-, 24-, and 30-months after start of trial
  Proportion of Hispanic patients who were successfully contacted for whom each mandatory component of enhanced care navigation was delivered
Order Printed PT Education Materials | 12-, 18-, 24-, and 30-months after start of trial
  Proportion of Hispanic patients with a new or existing spine pain problem who receive an auto-order for physical therapy education materials printed with the after visit summary at index encounter
Order Portal PT Education Materials | 12-, 18-, 24-, and 30-months after start of trial
  Proportion of Hispanic patients referred to physical therapy who receive an auto-order for electronic physical therapy education materials, referral information, and educational video in the patient portal
Order Text PT Education Materials | 12-, 18-, 24-, and 30-months after start of trial
  Proportion of Hispanic patients referred to physical therapy who are sent an auto-order for text link to physical therapy referral information and education video
Patient Portal Views | 12-, 18-, 24-, and 30-months after start of trial
  Proportion of Hispanic patients referred to physical therapy who view electronic physical therapy education materials, referral information, and education video from links provided in patient portal
Patient Text Views | 12-, 18-, 24-, and 30-months after start of trial
  Proportion of Hispanic patients referred to physical therapy who view physical therapy referral information and education video from links provided from the auto-text message

CONTACTS AND LOCATIONS:
Overall Officials: Katrina Monroe, PT, PhD, Principal Investigator — San Diego State University; Sara Gombatto, PT, PhD, Principal Investigator — San Diego State University Research Foundation
Locations (1):
- Family Health Centers of San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying published results will be shared via the Open Science Framework (OSF) repository, along with the study protocol, data dictionaries, statistical analysis plan, and intervention materials.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available beginning 12 months after publication of primary results and for a period of 5 years thereafter.
Access Criteria: Researchers must submit a written request and scientific justification for access to IPD and provide a data use agreement outlining compliance with confidentiality and ethical standards. Requests will be reviewed by the multiple principal investigator team and the FQHC research oversight committee. If approved, access will be granted through permissions in the Open Science Framework repository. Supporting materials will include the study protocol, data dictionaries, statistical analysis plan, and intervention materials.